CLINICAL TRIAL: NCT04321902
Title: Results of Surgical Management According to the Type of Empirical Antibiotics in Acute Inflammatory Gallbladder Disease; a Randomized Controlled Trial
Brief Title: Empirical Antibiotics in Acute Inflammatory Gallbladder Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul St. Mary's Hospital (Other)
Responsible Party: Principal Investigator, Taeho Hong, Professor, Seoul St. Mary's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Seoul-08
Record Dates: First submitted 2019-07-16; First posted 2020-03-25 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Cholecystitis, Acute
Keywords: empirical antibiotics; postoperative complication
MeSH Terms: conditions — Cholecystitis, Acute; Postoperative Complications | interventions — Cholecystectomy, Laparoscopic; Hematologic Tests; Blood Chemical Analysis; Urination; Blood Coagulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The experimental group in acute cholecystitis (Experimental): inclusion criteria
  1. among patients with mild acute cholecystitis (grade I by Tokyo guidelines) or moderate acute cholecystitis without evidence of gallbladder perforation(grade II)
  2. cholecystitis with a thickness of 4 mm or more on gallbladder in preoperative imaging
  3. Gallbladder with surrounding organs due to gallbladder inflammation
  4. Patients over 19 years of age
  First-generation cephalosporin (Cefazolin inj., 1g, Cefazolin sodium, Chong-geun-dang pharm.co.) was used as before and during surgery.
  Interventions: Procedure: Laparoscopic cholecystectomy
- The controled group in acute cholecystitis (Experimental): 1. among patients with mild acute cholecystitis (grade I by Tokyo guidelines) or moderate acute cholecystitis without evidence of gallbladder perforation(grade II)
  2. cholecystitis with a thickness of 4 mm or more on gallbladder in preoperative imaging
  3. Gallbladder with surrounding organs due to gallbladder inflammation
  4. Patients over 19 years of age
  Sencond-generation cephalosporin (Shincef inj., 750mg, Cefuroxime sodium, Shin-poong pharm.co.) was used as before and during surgery.
  Interventions: Procedure: Laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: Laparoscopic cholecystectomy — Method of operation
  1. Surgery was started under general anesthesia
  2. A trocar of 10 mm was placed on the navel, 5 mm under the blade, and 5 mm trocar was placed on the right upper abdomen.
  3. Pneumoperitoneum was performed using CO2 gas in the abdominal cavity.
  4. Dissection started from Calot's triangle and the operation was performed by retrograde cholecystectomy.
  5. The excised gallbladder was placed in a laparoscopic pocket and extracted through the umbilicus.
  6. The trocar was removed and the skin was sutured
  On the 1st day after surgery, hematology, blood chemistry, urine, blood clotting, and chest x-rays were performed. (Inspection and treatment were performed according to the current clinical pathway of gallbladder surgery)
  Other Names: hematology, blood chemistry, urine, blood clotting, and chest x-rays were performed

SUMMARY:
In this study, the investigators compared the surgical outcomes according to the type of antibiotics before surgery in patients who did not have evidence of systemic infection during acute cholecystitis.

The primary purpose of the study was to determine the type of preoperative antibiotics in patients who were scheduled for cholecystectomy, because of the mild (grade I) or moderate (grade 2) acute inflammatory gallbladder disease without gallbladder perforation. The investigators compared the incidence of postoperative complications according to the types of preoperative antibiotics(the first-generation vs second-generation cephalosporin).

The secondary purpose of the study was to confirm the clinical efficacy of first-generation cephalosporins following the use of empirical antibiotics. And the investigators compare with postoperative pain, postoperative hospital stay, re-hospitalization, and need for additional treatment. In addition, the investigators compare the postoperative complications, such as atelectasis and postoperative ileus.

DETAILED DESCRIPTION:
1. Background In the case of acute cholecystitis, in which acute inflammation was manifested in patients with gallstones and was accompanied by pain and fever, cholecystectomy through surgery was the standard treatment, and the use of empirical antibiotics to treat inflammation and prevent exacerbation until surgery was performed It was essential. However, as to which antibiotics were used as empirical antibiotics before cholecystectomy among various types of antibiotics, a variety of first-generation cephalosporins or second-generation cephalosporins had been selected and used depending on the existing practice or a physician's supervision. There was insufficient objective research and rationale for the selection of these empirical antibiotics. In addition, the use of high-grade antibiotics that are not required (eg, second-generation cephalosporins) might lead to prolonged hospital stays, wasted medical resources, increased medical expenses, and the occurrence of multi-drug resistant bacteria. In fact, the second-generation cephalosporin antibiotics had a price that was about two to four times higher depending on the product than the first-generation cephalosporin antibiotics. Therefore, in the use of empirical antibiotics before surgery for acute inflammatory gallbladder disease, if the same anti-inflammatory effect and postoperative results could be obtained with the first-generation cephalosporin antibiotics, there was no need to use expensive high-grade antibiotics required as empirical antibiotics before surgery. Moreover, side effects which could caused by high-grade antibiotics would be prevented.

   Therefore, in this study, the investigators tried to determine the effective and rational type of empirical antibiotics through random comparison experiments of two groups of patients according to the type of empirical antibiotics used in laparoscopic surgery in patients with acute cholecystitis without evidence of systemic infection. In addition, a double-blind prospective randomized control study comparing the first-generation and second-generation cephalosporin antibiotics commonly used in practice in clinical practice had not been published in Korea, and its clinical usefulness was expected to be great.
2. Code name of clinical trial drug or medical device or generic name of main ingredient, raw material drug (raw material in case of medical device) and its quantity, formulation (form / structure / number in case of medical device), etc.

<!-- -->

1. Test drug ; Cefazolin inj., 1 g, Cefazolin sodium, white crystal, vial injection with crystalline powder or lump
2. control drug ; Shincef inj., 750mg, Cefuroxime sodium, colorless transparent vial injection with light yellow powder

3. Target disease Acute cholecystitis without evidence of gallbladder perforation among mild (Grade I) and severe (Grade II) classification of acute cholecystitis according to Tokyo guidelines

4. Subject selection criteria, exclusion criteria, number of target subjects and their rationale <Inclusion criteria>

1. among patients with mild acute cholecystitis (grade I by Tokyo guidelines) or moderate acute cholecystitis without evidence of gallbladder perforation(grade II)
2. cholecystitis with a thickness of 4 mm or more on gallbladder in preoperative imaging
3. Gallbladder with surrounding organs due to gallbladder inflammation
4. Patients over 19 years of age <Exclusion criteria>

1) patients with elective gallbladder surgery (chronic cholecystitis) 2) gallbladder disease not inflammatory disease (GB cancer, GB polyp) 3) pregnant women, patients under 18 years of age, over 70 years of age 4) patients with simultaneous surgery due to other organ diseases 5) immunosuppressed patients; liver transplant patients, kidney transplant patients, acquired immunodeficiency syndrome patients 6) patients with hemorrhagic tendency, or with hematologic diseases 7) Patients who underwent percutaneous cholecystectomy (PTGBD) 8) Patients with acute cholecystitis who had gallbladder perforation, grade II or III by Tokyo guidelines 9) Drain tube is required during surgery (eg. if delayed biliary leakage was concerned, hepatic duct injury was suspected or cystic duct ligation was incomplete during operation.) <Calculation and basis of the number of target subjects> In the previous studies, infectious complications after laparoscopic surgery for acute inflammatory gallbladder disease have been reported as 18.5%. The investigators designed a non-inferiority test (non-inferiority limit of 13%) assuming postoperative infectious complication of 18.5% confidence level of 95%, and assigned 167 to each group considering the dropout rate of 10%

5. Random allocation schedule and operation Randomization was performed using block randomization without stratification, and a block size of 2, 4 or 6 was applied to complete the randomization table to maintain unpredictability, which was the basic principle of randomization. .

Assignment bags with random assignment numbers and assigned groups were made of opaque material so that they could be blinded and remain sealed until random assignment was performed for each subject.

The person in charge of the clinical trial or the person in charge of the clinical trial finally checked the exclusion criteria and, if it was a suitable subject, a random number was assigned and stored in the allocation bag. Thereafter, the management pharmacist receives the assignment bag with the assignment number, releases the seal of the assignment bag, and prescribes antibiotics according to the administration group assigned to the subject according to each random assignment number. Afterwards, the managed pharmacist brought the antibiotics according to the newly developed drug code for the clinical trial in accordance with the [Medical Clinical Trial Management Standards (related to Article 30, Paragraph 1)], and then administered to the patient. The management pharmacist should record the release information (release date and releaser) immediately after the release of the assignment bag which the random assignment enveloped, when it had already been released once, it could not reassign the randomization code to other subjects even if the subject withdraws consent.

6. Clinical trial period clinical trial approval date-2021-04-30

7. Clinical trial method (administration / dosage, administration / use method, administration / use period, combination therapy, etc.)

1. Research Design Prospective randomized controlled trial in two groups
2. Describe what treatment is performed for the experimental group / control group A. Clinical trial flow

<!-- -->

1. Before the patient's surgery, hematology, blood chemistry, blood coagulation, urine, Chest X-ray, EKG, and Abdomen CT were performed in accordance with current clinical practice guidelines.
2. Select the patient group that met the diagnostic criteria according to the test results above.
3. Select a random patient group to determine the type of empirical antibiotic to use before surgery
4. For each selected group, intravenous antibiotics (Cefazolin inj., 1 g, Cefazolin sodium versus. Shincef inj., 750 mg, Cefuroxime sodium) were used as before and during surgery.

   - The clinical trial manager or the clinical trial manager finally checked the criteria for selection exclusion and, if it was a suitable subject, a random number was assigned and stored in the allocation bag. Thereafter, the management pharmacist received the assignment bag with the assignment number, released the seal of the assignment bag, and prescribed antibiotics according to the administration group assigned to the subject according to each random assignment number. Afterwards, the managed pharmacist brought the antibiotics according to the newly developed drug code for the clinical trial in accordance with the [Medical Clinical Trial Management Standards (related to Article 30, Paragraph 1)], and then administered to the patient.
5. After surgery, both groups were discharged through the same recovery process after surgery.
6. On the 1st day after surgery, hematology, blood chemistry, urine, blood clotting, and chest x-rays were performed. (Inspection and treatment were performed according to the current clinical pathway of gallbladder surgery)
7. If there are no specifics, a fluid diet was performed starting from lunch on the first day after surgery.
8. If there were no specifics, patient would be discharged on the second day after surgery.
9. Stability and effectiveness were monitored during hospitalization and after discharge.

B. Method of operation

1. Surgery was started under general anesthesia
2. A trocar of 10 mm was placed on the navel, 5 mm under the blade, and 5 mm trocar was placed on the right upper abdomen.
3. Pneumoperitoneum was performed using CO2 gas in the abdominal cavity.

   * Double pressure through CO2 gas was maintained at 12mmHg / and 2L / min.
4. Dissection started from Calot's triangle and the operation was performed by retrograde cholecystectomy.

   * The cystic duct was ligated with a 10mm clip and the cystic artery was ligated with a 10mm clip as well.
   * If the cystic duct was unstablely ligated, ligation was performed through an endoloop.
   * After ligation, the gallbladder was dissected from the liver.
5. Washed the surgical site.
6. The excised gallbladder was placed in a laparoscopic pocket and extracted through the umbilicus.
7. The trocar was removed, the skin was sutured, and the operation was completed. C. Discharge Principle

<!-- -->

1. When hematologically stable and vital signs were stable
2. When the patient's condition was stable by proceeding to the normal diet

8. characteristics of observational and clinical test <Observation test>

1) Medical history investigation Before entering the clinical trial, checked the following items through interviews, chart and questions about the subject's background (demographic information), medical history, etc., and recorded them in the record.

1. Background investigation: Subject's initials, date of birth, sex, feasibility of pregnancy, pregnancy, lactation
2. medical history
3. History history: History of other diseases 2) Physical examination, vital signs examination Investigators checked whether the body organs were normal or abnormal through medical examination and examination and any significant findings found during the examination should be recorded in the physical examination column of the record sheet, and confirmed to be suitable for participation in the study.

After surgery, the pain level was measured by questioning the patient himself using the VAS score, and the amount of analgesics (injection drugs; tramadol and oral drugs; ircodon) administered after surgery to the patient was recorded through medication records.

3) Clinical examination

It was performed during the hospitalization after decision to perform cholecystectomy. Blood sampling for the subjects was performed aseptically. Investigators recorded the test results, determined whether they were normal or abnormal, and record the opinions of researchers regarding abnormal values. Clinical tests included :

1. Hematology tests: Hematocrit, Hemoglobin, MCV, MCH, MCHC, Platelet, WBC & Differential count, ESR
2. Blood coagulation test: PT INR, aPTT, BT
3. Blood chemistry test: SGOT (AST), SGPT (ALT), alkaline phosphatase, γ-GTP, bilirubin (total / direct), fasting plasma glucose, BUN, creatinine, sodium, potassium, chloride, calcium, phosphorus, magnesium , total protein, albumin, uric acid, CPK, LDH, free fatty acid, CRP, HbA1c, CRP
4. Urine test: Color, specific gravity, pH, Leucocytes, Nitrite, Protein, Glucose, Ketone, Urobilinogen, Bilirubin, Microscopy (RBC, WBC) 4) Imaging medical examination

<!-- -->

1. Before surgery, chest X-ray and electrocardiography were performed to evaluate whether surgery was possible.
2. Imaging studies such as CT, Sonogram, and MRCP were conducted. 5) Postoperative hospital stay The day after surgery, hematology, blood chemistry, urine, blood clotting, Chest x-ray.

6) Check for infection.

* Surgical site infection

  1. Confirmation at every patient visit. Troca insertion site was defined as superficial surgical site infection if there was redness, heat sensation and abscess.
  2. If there was fluid retention and abscess around the surgical site in the abdominal cavity, it was defined as deep surgical site infection.
* Distant infection

  * Respiratory, urinary system infections and bacteremia or lymphangitis 7) Check for leakage of bile.
* Groups who had drainage catheter would be checked through the drainage pattern. In the group without drainage catheter, after surgery, if there is epigastric pain, indigestion, fever, and jaundice, a selective medical imaging test (CT, sonogram, MRCP) was performed.

  8) Surgery time, bleeding amount were described. 9) Postoperative complications (things other than those described above) were described.

  9. Predicted side effects and precautions

  1) Side effects that might occur in the experimental group (the first-generation cephalosporin use group)
* Wound infections and deep infections : Since antibiotics were used, the possibility was very low.
* Side effects of antibiotics (allergic reaction) 2) Side effects that could be occurred in the control group (2nd generation cephalosporin use group)
* Extension of the period of stay
* Increased hospitalization costs
* Increase of multi-drug resistant bacteria
* Side effects of antibiotics (allergic reaction) (In the event of side effects, medical judgment was used to actively select a therapeutic method.)

  10. Stop or drop the test Dosing and testing should be discontinued if any of the following occurs, and the reasons for discontinuation and findings should be recorded.
  1. After surgery, when a side effect that was life-threatening, the investigator determined that it was necessary to stop
  2. When the patient refused or withdrew consent after starting the test
  3. If the patient was inadequate after starting the test
  4. After the start of the test, if patient had received treatment that might affect the course of treatment, such as other combination drugs and herbal treatments, without the permission of the test manager
  5. After the start of the test, it was judged that it was impossible to conduct inspection or investigation due to the circumstances
  6. After surgery, when surgery was required due to a disease of another organ not related to gallbladder surgery.

  11. Statistical analysis
  1. Analysis of validity variables A. Analysis of primary efficacy variables.

     * During the postoperative hospital stay, the incidence of wound infection and deep infection rates in the group using the first-generation cephalosporin and the second-generation cephalosporin as an empirical antibiotic before surgery was determined by the student's t-test or according to the satisfaction of the normal distribution assumption. Test using wilcoxn's rank sum test, and present the descriptive statistics (average, standard deviation, median, minimum, and maximum). Also, the difference in the incidence of infection between the two groups (test group-control group) was presented as the mean and 95% confidence interval, and if it was less than the non-inferiority limit of 13%, the group using the first-generation cephalosporin antibiotics was the second-generation cephalosporin. It was not inferior to the group using antibiotics. That was, it would decide that it was not inferior.

     B. Complications after surgery.
     * Complications will be defined and analyzed through researchers' experience and review of existing literature.

       * Fever after surgery: Fever of 37.5 ° C or more that lasts at least 48 hours after surgery.

         * Surgical site infection: In case of seroma, hematoma, or abscess in the surgical incision.

           * Surgery wound wound: When the wound was opened and opened. ④ Coming, vomiting after surgery: If patient needed to use antiemetic after 24 hours of surgery, or if patient had vomited even once.

             * Sustained shoulder pain after surgery: If patient complained of a stiff shoulder until the outpatient follow-up examination (one week after discharge).

               ⑥ Bleeding after surgery: When the patient's vital signs change or there was a decrease in Hb 2.0 or higher on the hemoglobin test the day after surgery.

               ⑦ Abscess in the abdominal cavity after surgery: When an abscess in the abdominal cavity was confirmed by image examination (ultrasound, CT, etc.) accompanied by fever and pain in the physical examination.

               ⑧ Persistent bowel obstruction: If the meal could not be started even after 2 days of surgery.
  2. Analysis of secondary efficacy variables In the case of categorical variables for the length of stay, surgical time, and complication data obtained as secondary endpoints, n (%) was presented, and the ratio difference between the two groups was tested using Chi-square or Fisher's exact test. In addition, for continuous variables, the mean, standard deviation, median, minimum, and maximum values were presented, and the normality test was performed to test with Student's t-test for normal distribution, and for the non-normal distribution, Wilcoxon rank-sum test The difference between the two groups would be tested. All statistical analysis would use SPSS version 21.0, and it would be judged that it was statistically significant below the significance level of 0.05.
  3. Analysis target group

  <!-- -->

  1. intention to treat analysis group Randomization would be performed only if the selection criteria described above were met, and all randomized subjects would be included in statistical analysis.
  2. per protocol analysis group The Per protocol analysis group was defined as a patient who had undergone randomization and had undergone chest imaging the next day after surgery, and whose pain had been assessed.

  4) How to deal with missing values This study was a prospective study, and it was expected that there would be no missing values of the main or secondary endpoints during the experiment. However, if a missing value occurred, the missing value was substituted with the average value.

  5) How to deal with compliance Since the intervention applied to this study was an intervention performed during surgery while the patient had general anesthesia, there would be no difference in treatment compliance. In addition, postoperative thoracic imaging and pain assessment were also included in the clinical pathway for laparoscopic cholecystectomy, so there was no difference in treatment compliance.

  12. Safety evaluation of side effects and reporting method In the event of adverse reactions and adverse reactions after surgery, trained the subject to report to the researcher, checked and recorded the occurrence of adverse reactions at each visit, symptoms, appearance time, duration, severity of adverse reactions, and causal relationship with the test drug Record in the report. In the event of a serious adverse event or unexpected problem, the responsible researcher should report it to the clinical trial.

  13. Compensation Protocol of victim Laparoscopic cholecystectomy was a safe operation with a very low risk of surgery. Also, there are basically no additional risks accompanying the study. Antibiotics were drugs that had been used before, so there are no additional complications beyond the known complications. If patient got injury or illness by participating in this study, medical treatment would be provided. In order to receive medical treatment related to the clinical symptoms or signs, investigators would make a quick diagnosis and receive treatment when needed through consultation.

ELIGIBILITY:
Inclusion Criteria:

1. among patients with mild acute cholecystitis (grade I by Tokyo guidelines) or moderate acute cholecystitis without evidence of gallbladder perforation(grade II)
2. cholecystitis with a thickness of 4 mm or more on gallbladder in preoperative imaging
3. Gallbladder with surrounding organs due to gallbladder inflammation
4. Patients over 19 years of age, under 70 years of age

Exclusion Criteria:

1. patients with elective gallbladder surgery (chronic cholecystitis)
2. gallbladder disease not inflammatory disease (GB cancer, GB polyp)
3. pregnant women, patients under 18 years of age, over 70 years of age
4. patients with simultaneous surgery due to other organ diseases
5. immunosuppressed patients; liver transplant patients, kidney transplant patients, acquired immunodeficiency syndrome patients
6. patients with hemorrhagic tendency, or with hematologic diseases
7. Patients who underwent percutaneous cholecystectomy (PTGBD)
8. Patients with acute cholecystitis who had gallbladder perforation, grade II or III by Tokyo guidelines

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2020-04-02 (Estimated); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Infectious Postoperative Complications | 30 days
  Incidence of infectious postoperative complications in patients who underwent a laparoscopic cholecystectomy due to grade I Tokyo guidelines for acute cholecystitis or grade II Tokyo guidelines for acute cholecystitis except the evidence of gallbladder perforation, with the first-generation cephalosporin and the second-generation cephalosporin.

SECONDARY OUTCOMES:
Duration of hospitalization | Participants will be followed for the duration of hospital stay, an expected average of 2 days
  The duration between the operation day and the day of discharge

CONTACTS AND LOCATIONS:
Overall Officials: Sung eun Park, MD, Study Director — The Catholic University of Korea
Locations (1):
- Department of HBP Surgery, Seoul St. Mary's hospital, Seoul, Seocho-gu, Banopo-dong, South Korea

IPD SHARING:
Plan to Share IPD: No